CLINICAL TRIAL: NCT06573307
Title: To Develop a Prognostic Model for Predicting Survival and Treatment Response for Advanced Gastric Cancer Patients After Neoadjuvant Therapy by Analyzing Hematological Markers Dynamic Load
Brief Title: Hematological Dynamic Scores for Predicting Survival and Treatment Response for Advanced Gastric Cancer After Neoadjuvant Therapy
Status: Completed | Type: Observational
Sponsor: Chang-Ming Huang, Prof. (Other)
Responsible Party: Sponsor-Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Organization: Fujian Medical University (Other)
Other Study IDs: FMUUH-0323
Record Dates: First submitted 2024-08-26; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Neoadjuvant chemotherapy; inflammation; Oxidative stress; Treatment response; Risk stratification
MeSH Terms: conditions — Stomach Neoplasms; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
HMDLS, based on hematological markers, could effectively distinguish the long-term efficacy of AGC patients after NAT. The predictive performance of nomogram-HMDLS was better than ypTNM stage, achieving better prognostic stratification and tumor treatment response prediction.

DETAILED DESCRIPTION:
In this research, we incorporated a total of 320 patients from the Union Hospital of Fujian Medical University to form the training cohort (TC). Additionally, we included 122 patients from four distinct medical centers to serve as the external validation cohort (EVC). The Hematological Marker Dynamic Load (ΔHMDL) was determined using the following formula: ΔHMDL = (HMDL pre-surgery - HMDL pre-NAT) / HMDL pre-NAT, where HMDL represents the hematological marker levels before surgery and before the initiation of Neoadjuvant Therapy (NAT), respectively.

Employing LASSO regression analysis, we identified the most influential and statistically significant ΔHMDL indicators. These were then utilized to compute the Hematological Marker Dynamic Load Score (HMDLS), defined as: HMDLS = Σ(LASSO coefficient * ΔHMDL), where the summation encompasses the products of the LASSO-estimated coefficients and the corresponding ΔHMDL values.

Further, leveraging the outcomes of a multivariate COX regression analysis, we integrated clinical parameters with the HMDLS to formulate a predictive model, termed the Nomogram-HMDLS model. The efficacy of this model in terms of predictive accuracy, clinical utility, and calibration was meticulously assessed and confirmed through several metrics, including the concordance index (C-index), Receiver Operating Characteristic (ROC) curve analysis, decision curve analysis (DCA), and calibration curves.

ELIGIBILITY:
Inclusion Criteria:

* (1) AGC with clinical stage T2-4NxM0 (cT2-4NxM0) before NAT, (2) no history of other malignant tumors, distant metastases or invasion of adjacent organs, and (3) patients who underwent radical gastrectomy after receiving NAT.

Exclusion Criteria:

* (1) history of upper abdominal surgery (except for the laparoscopic cholecystectomy), (2) history of upper abdominal radiotherapy, (3) emergency surgery, or palliative surgery, (4) continuous use of medications such as anticoagulant, antiplatelet, and leukocyte-boosting drugs that significantly affect hematological markers during therapy, and (5) incomplete clinical and follow-up data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In this study, we retrospectively collected clinicopathologic data and hematological markers before Neoadjuvant therapy and surgery in AGC patients who had undergone Neoadjuvant therapy and received radical gastrectomy in five hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 442 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
3-year OS | 3-year OS or 36 months
  Overall survival, death, survival with tumor
3-year DFS | 3 years DFS or 36 months
  Disease-free survival, death,recurrence
Tumor Regression Grade | 3 years or 36 months
  a grade system evaluates the pathological response based on the degree of tumor tissue regression after NAT.

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Department of Gastric Surgery， Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No